CLINICAL TRIAL: NCT06754397
Title: Diagnostic Accuracy of Magnetic Resonance Cholangiopancreatography as Compared to Ultrasound and Computed Tomography in Patients With Obstructive Jaundice
Brief Title: Diagnostic Accuracy of Magnetic Resonance Cholangiopancreatography in Patients With Obstructive Jaundice
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Demiana Mohsen Soliman, Radiological resident, Sohag University
Other Study IDs: Soh-Med--24-12-04MS
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Obstructive Jaundice
MeSH Terms: conditions — Jaundice, Obstructive | interventions — Cholangiopancreatography, Magnetic Resonance; Ultrasonography; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with obstructive jaundice: MRCP as a role that is used as a non-invasive diagnostic tool for visualizing the pancreaticobiliary tree without the use of contrast media
  Interventions: Diagnostic Test: Magnetic Resonance Cholangiopancreatography

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Cholangiopancreatography — Three most important sequences included axial T2 weighted scan from liver to ampullary region followed by T2 weighted 3D FSE sequence acquired in coronal oblique plane using respiratory triggering by tying bellows over abdomen. After this breath hold HASTE sequence is acquired in coronal plane. Maximum intensity projection (MIP) and thick slab images are also used for interpretation. US, CECT and MRCP scans are interpreted by radiologists blinded to other imaging findings
  Other Names: Ultrasound; Computed tomography

SUMMARY:
Evaluate the diagnostic accuracy of Magnetic Resonance Cholangiopancreatography (MRCP) compared with Ultrasound and Computed Tomography (CT) in patients with obstructive jaundice taking findings of ERCP/ PTC and histopathology as gold standard.

DETAILED DESCRIPTION:
MRCP as a diagnostic role to determine the presence and severity of biliary and pancreatic ductal dilatation. It can also detect the length of the stricture as well as the exact cause and location of the obstructing lesion in comparison to other modalities.

ELIGIBILITY:
Inclusion Criteria:

Adult male and female patients clinically diagnosed obstructive jaundice are included in the study with positive laboratory tests.

Exclusion Criteria:

Patients with non-obstructive (prehepatic/hepatic) cause of jaundice. Patients having contraindications to perform MRI (Patients with any electrically, magnetically or mechanically activated implants, pacemaker, cochlear implants or any metallic orthopedic implants and claustrophobic patients).

Ages: 15 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult male and female patients clinically diagnosed obstructive jaundice are included in the study with positive laboratory tests.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of Magnetic Resonance Cholangiopancreatography in patients with obstructive jaundice according to the findings | Within twelve months
  Magnetic Resonance Cholangiopancreatography findings in patients with obstructive jaundice comparing to findings of ERCP/ PTC and histopathology .

CONTACTS AND LOCATIONS:
Overall Officials: Magdy M Amin, Professor, Study Director — Medical research ethics committee - Sohag university

IPD SHARING:
Plan to Share IPD: Undecided